CLINICAL TRIAL: NCT01549886
Title: A Randomized, Open-Label, Multi-Center, Phase 2 Study of Zevalin ([90Y]- Ibritumomab Tiuxetan) Versus Zevalin and Motexafin Gadolinium in Patients With Rituximab- Refractory Low-grade or Follicular B-cell Non-Hodgkin's Lymphoma
Brief Title: Phase 2 Study of Zevalin Versus Zevalin and Motexafin Gadolinium in Patients With Rituximab-Refractory Low-grade or Follicular B-cell Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to business reasons.
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPI-MGD-11-201
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Results first posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Zevalin; Motexafin Gadolinium
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — ibritumomab tiuxetan; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MGD + Rituximab + Y-90-Zevalin (Experimental): Moxtezafin Gadolinium: Day 1-4 Motexafin gadolinium 5 mg/kg intravenously once daily, followed in one hour (Day 1 only) by Day 1 Rituximab 250 mg/m^2 intravenous infusion.
  Day 8-11 Motexafin gadolinium 5 mg/kg intravenously once daily, followed in one hour (Day 8 only) by Day 8 Rituximab 250 mg/m^2 intravenous infusion, followed 4 hours later by Y-90-Zevalin 0.4 millicurie / kilogram (mCi/kg) 10-minute intravenous push (0.3 mCi/kg in patients with a platelet count in 100,000/μL to 149,000/μL.
  Interventions: Drug: Y-90-Zevalin; Drug: Moxtezafin Gadolinium; Drug: Rituximab
- Rituximab + Y-90-Zevalin (Active Comparator): Day 1 Rituximab 250 mg/m^2 intravenous infusion. Day 8 Rituximab 250 mg/m^2 intravenous infusion, followed 4 hours later by Y-90-Zevalin 0.4 mCi/kg 10-minute intravenous push
  Interventions: Drug: Y-90-Zevalin; Drug: Rituximab

INTERVENTIONS:
Drug: Y-90-Zevalin — Day 8 - Y-90-Zevalin 0.4 mCi/kg 10-minute intravenous push
  Other Names: [90Y]- ibritumomab tiuxetan (Zevalin)
Drug: Moxtezafin Gadolinium — Day 1-4 Motexafin gadolinium 5 mg/kg intravenously once daily, followed in one hour (Day 1 only) by Day 1 Rituximab 250 mg/m^2 intravenous infusion.
  Day 8-11 Motexafin gadolinium 5 mg/kg intravenously once daily
  Other Names: MGD
  Arms: MGD + Rituximab + Y-90-Zevalin
Drug: Rituximab — Day 1 and Day 8: Rituximab 250 mg/m^2 intravenous infusion

SUMMARY:
The objectives of this study are to evaluate the efficacy and safety of the Zevalin regimen compared to Zevalin and motexafin gadolinium in patients with rituximab-refractory, low-grade or follicular Non-Hodgkin's Lymphoma (NHL).

Effectiveness of the experimental regimen assessed by complete response rate within 6 months of study entry (primary endpoint), complete response rate within 3 months of study entry, and overall response rate within 6 month of study entry.

DETAILED DESCRIPTION:
This multi-center, randomized, open-label study is designed to compare the safety and efficacy of therapy with Zevalin regimen versus Zevalin and motexafin gadolinium in patients with rituximab-refractory, low-grade or follicular NHL. Approximately 100 adult patients enrolled in the study (approximately 50 in each group at 15 clinical sites in North America).

Patients screened for eligibility within the 14 days prior to Day 1 of the study. Once written informed consent has been obtained and patient eligibility has been established, the patient randomized 1:1 to receive either Zevalin or Zevalin and motexafin gadolinium.

Patients assessed for safety at each visit to the study center and for disease response at Months 3, 6 and 12. An end-of-study-visit performed at Month 12.

Disease status assessed using positron emission tomography (PET) or PET/computerized tomography (CT), and/or flow cytometry. Disease response will be evaluated in accordance with the standardized definitions and criteria of the International Working Group Revised Response Criteria for Malignant Lymphoma. The efficacy endpoints that assessed are complete response rate and overall response rate.

Safety was assessed by adverse events, physical examinations, vital signs, and clinical laboratory assessments. Serious adverse events (SAEs) and treatment-emergent adverse events (TEAEs) was collected for all patients beginning on Day 1 and continuing through the end-of study-visit to be performed at Month 12 or withdrawal from study.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, at least 18 years of age
2. Histologically-confirmed follicular or indolent, marginal zone and small lymphocytic B cell non-Hodgkin's lymphoma
3. Progressive disease within 6 months of the end of a rituximab-containing regimen; or progressive disease at any time following 2 or more prior rituximab-containing regimens; or progressive disease while on rituximab-containing regimen.
4. At least 1 measurable tumor (> 1.5 cm in the long axis and > 1.0 cm in the short axis) that has not been irradiated previously or that has increased in size since previous irradiation
5. A life expectancy of at least 3 months
6. A World Health Organization/Eastern Cooperative Oncology Group (WHO/ECOG) performance status of 0 or 1
7. Adequate hematopoietic function: absolute neutrophil count (ANC) ≥ 1,500 cells/μL, absolute lymphocyte count (ALC) ≤ 5,000 cells/μL, platelet count ≥ 100,000 cells/μL,hemoglobin ≥ 9 g/dL (may be transfused to maintain this concentration). Patients who have received pre-phase therapy for purposes of improving performance status prior to initiating Zevalin are eligible.
8. Adequate liver function: total bilirubin ≤ 2 × upper limit of normal (ULN), Aspartate aminotransferase (AST) (Serum glutamic oxaloacetic transaminase [SGOT]) and Alanine transaminase (ALT) (Serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 × upper limits of normal (ULN)
9. Creatinine clearance ≥ 60 mL/min/1.73 m^2
10. Bone marrow involvement < 25%
11. If men or women of reproductive potential, agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for at least 1 year following treatment with Zevalin
12. Willing and able to provide written Informed Consent and to comply with the requirements of the study protocol

Exclusion Criteria:

1. Received antineoplastic, experimental, and/or radiation therapy within the 3 weeks prior to Study Day 1
2. Has not recovered to ≤ Grade 1 from all toxicities related to prior treatments
3. Prior radioimmunotherapy for NHL
4. Autologous stem cell transplant within the 3 months prior to Study Day 1, and/or any history of allogeneic stem cell transplant with continued allogeneic hematopoiesis
5. Platelet transfusion within the 7 days prior to Study Day 1
6. History of porphyria
7. Grade 2 or higher peripheral neuropathy within the 14 days prior to Study Day 1
8. History of or active central nervous system disease (e.g., primary brain tumor, seizures not controlled with standard medical therapy, brain metastases)
9. Ongoing, active infection that requires anti infective therapy
10. Clinically significant cardiovascular disease (e.g., unstable angina pectoris, serious cardiac arrhythmia requiring medication, uncontrolled hypertension, myocardial infarction, New York Heart Association [NYHA] Class 2 or higher congestive heart failure, Grade 2 or higher peripheral vascular disease) within the 12 months prior to Study Day 1
11. History of another clinically significant medical condition, metabolic dysfunction, physical examination finding, and/or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or place the patient at high risk of treatment complications and/or of noncompliance with the study procedures
12. Major surgical procedure and/or significant traumatic injury (that which could interfere with the patient's ability to receive protocol therapy as determined by the principal investigator) within the 28 days prior to Study Day 1, and/or patient is anticipated to require a major surgical procedure during the study period
13. Diagnosed with and/or treated for a malignancy other than NHL within the 2 years prior to Study Day 1, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, and/or low-risk prostate cancer after curative therapy from which the patient has been disease-free for at least 1 year
14. Evidence of a bleeding diathesis and/or a coagulopathy
15. Known HIV infection
16. Known hypersensitivity to drugs with porfyrin-like structures, like Visudyne™.
17. Positive Hepatitis B or C infection: Patient must be tested for hepatitis B surface antigen.
18. Pregnant or lactating woman
19. Full dose oral or parenteral anticoagulants within the 10 days prior to Study Day 1, and/or anticipated full dose oral or parenteral anticoagulant therapy during the study period(except as required to maintain patency of pre-existing, permanent, indwelling intravenous catheters) or thrombolytic agents
20. Participated in another clinical study within the 4 weeks prior to Study Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Evens, DO, MSc, Principal Investigator — University of Massachusetts, Worcester
Locations (9):
- United States (9):
  - Alta Bates Summit Medical Center-Herrick, Berkeley, California
  - Providence Saint Joseph Medical Center, Burbank, California
  - Halifax Health- Center for Oncology, Daytona Beach, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Loyola University Chicago, Maywood, Illinois
  - Oncology Specialists, Park Ridge, Illinois
  - University of Massachusetts - Worcester, Worcester, Massachusetts
  - Hackensack Medical Center, Hackensack, New Jersey
  - West Virginia University, WVU Healthcare, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- MGD+Rituximab+Y-90-Zevalin: Moxtezafin Gadolinium: Day 1-4 Motexafin gadolinium 5 mg/kg intravenously once daily, followed in one hour (Day 1 only) by Day 1 Rituximab 250 mg/m^2 intravenous infusion.
  Day 8-11 Motexafin gadolinium 5 mg/kg intravenously once daily, followed in one hour (Day 8 only) by Day 8 Rituximab 250 mg/m^2 intravenous infusion, followed 4 hours later by Y-90-Zevalin 0.4 millicurie/kilogram (mCi/kg) 10-minute intravenous push (0.3 mCi/kg in patients with a platelet count in 100,000/μL to 149,000/μL.
- Rituximab+Y-90-Zevalin: Day 1 Rituximab 250 mg/m^2 intravenous infusion. Day 8 Rituximab 250 mg/m^2 intravenous infusion, followed 4 hours later by Y-90-Zevalin 0.4 mCi/kg 10-minute intravenous push (0.3 mCi/kg in patients with a platelet count in 100,000/μL to 149,000/μL.)
Period: Overall Study
Arm/Group | MGD+Rituximab+Y-90-Zevalin | Rituximab+Y-90-Zevalin
Started | 2 | 3
Completed | 0 | 0
Not Completed | 2 | 3
Not completed — Sponsor's decision | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- MGD+Rituximab+Zevalin: Moxtezafin Gadolinium: Day 1-4 Motexafin gadolinium 5 mg/kg intravenously once daily, followed in one hour (Day 1 only) by Day 1 Rituximab 250 mg/m^2 intravenous infusion.
  Day 8-11 Motexafin gadolinium 5 mg/kg intravenously once daily, followed in one hour (Day 8 only) by Day 8 Rituximab 250 mg/m^2 intravenous infusion, followed 4 hours later by Y-90-Zevalin 0.4 mCi/kg 10-minute intravenous push (0.3 mCi/kg in patients with a platelet count in 100,000/μL to 149,000/μL.
- Rituximab+Zevalin: Day 1 Rituximab 250 mg/m^2 intravenous infusion. Day 8 Rituximab 250 mg/m^2 intravenous infusion, followed 4 hours later by Y-90-Zevalin 0.4 mCi/kg 10-minute intravenous push (0.3 mCi/kg in patients with a platelet count in 100,000/μL to 149,000/μL.)
- Total: Total of all reporting groups
Arm/Group | MGD+Rituximab+Zevalin | Rituximab+Zevalin | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (2.5) | 57 (6.24) | 54 (4.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (CR)
Time Frame: 6 Months
Population: Data for this outcome measure was not collected and analysed as no participants available for analysis and study was discontinued prematurely due to business reasons.
Groups:
- MGD+Rituximab+Y-90-Zevalin: Moxtezafin Gadolinium: Day 1-4 Motexafin gadolinium 5 mg/kg intravenously once daily, followed in one hour (Day 1 only) by Day 1 Rituximab 250 mg/m2 intravenous infusion.
  Day 8-11 Motexafin gadolinium 5 mg/kg intravenously once daily, followed in one hour (Day 8 only) by Day 8 Rituximab 250 mg/m2 intravenous infusion, followed 4 hours later by Y-90-Zevalin 0.4 mCi/kg 10-minute intravenous push (0.3 mCi/kg in patients with a platelet count in 100,000/μL to 149,000/μL.
- Rituximab+Y-90-Zevalin: Day 1 Rituximab 250 mg/m2 intravenous infusion. Day 8 Rituximab 250 mg/m2 intravenous infusion, followed 4 hours later by Y-90-Zevalin 0.4 mCi/kg 10-minute intravenous push (0.3 mCi/kg in patients with a platelet count in 100,000/μL to 149,000/μL.)
  Zevalin Regimen: Day 1 - Rituximab 250 mg/m2 intravenous infusion. Day 8 - Rituximab 250 mg/m2 intravenous infusion, followed 4 hours later by Y-90-Zevalin 0.4 mCi/kg 10-minute intravenous push
Arm/Group | MGD+Rituximab+Y-90-Zevalin | Rituximab+Y-90-Zevalin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Response Rate
Description: Complete response rate within 3 months, overall response rate within 6 months and progression-free survival.
Time Frame: 3 Months and 6 Months
Population: as for outcome 1
Arm/Group | MGD+Rituximab+Zevalin | Rituximab+Zevalin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Serious Adverse Events and Non-Serious Adverse Events
Description: An Adverse Events (AE) was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly. Non-SAEs was an AE events that are not Serious Adverse Events.
Time Frame: From time of dosing until 2 years
Population: Safety analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | MGD+Rituximab+Y-90-Zevalin | Rituximab+Y-90-Zevalin
Number analyzed (Participants) | 2 | 3
Participants
  Serious Adverse Events | 1 | 2
  Non-Serious Adverse Events | 2 | 3

ADVERSE EVENTS:
Time Frame: AEs were collected from time of dosing until 2 years.
Arm/Group | MGD+Rituximab+Y-90-Zevalin | Rituximab+Y-90-Zevalin
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/3
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MGD+Rituximab+Y-90-Zevalin (N=2) | Rituximab+Y-90-Zevalin (N=3)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
UTI (Infections and infestations) | 0 (0) | 1 (1)
Thrombocytopenia (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MGD+Rituximab+Y-90-Zevalin (N=2) | Rituximab+Y-90-Zevalin (N=3)
Abdominal Discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neutrophils count decreased (Investigations) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No